CLINICAL TRIAL: NCT05891184
Title: Color Doppler Ultrasound and Transient Elestoghraphy as Predictors for Presence of Gastroesophageal Varices and Variceal Bleeding in Patients With Liver Cirrhosis
Brief Title: Color Doppler US and TE as Predictors for Presence of Gastroesophageal Varices and Variceal Bleeding in Patients With LC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham Mamdouh Kemaly, Waleed Attia, Hanan Nafeh, Assiut University
Other Study IDs: Dopper Us and TE in LC
Record Dates: First submitted 2023-05-26; First posted 2023-06-06 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Gastroesophageal Varices Hemorrhage
Keywords: color doppler ultrasound; transient elastography; liver cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Gastroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: the 1st group will be patients with current or past history of variceal bleeding,
  Interventions: Device: color doppler ultrasound, transient elastography, upper endoscopy
- 2: the 2nd group will be patients having gastroesophageal varices without variceal bleeding,
  Interventions: Device: color doppler ultrasound, transient elastography, upper endoscopy
- 3: 3ed group will be patients without gastroesophageal varices or variceal bleeding.
  Interventions: Device: color doppler ultrasound, transient elastography, upper endoscopy

INTERVENTIONS:
Device: color doppler ultrasound, transient elastography, upper endoscopy — Abdominal US: for detecting the portal hypertension, splenomegaly and portosystemic abdominal collaterals .
  Doppler US: detecting the diameter and mean blood flow velocity, blood flow volume, perfusion pressure gradient, congestion index, resistive index, pulsatility index of hepatic artery and platelet count-to-spleen diameter ratio will be performed using logic 10 with a 3.5-MHz duplex convex transducer, in supine position after overnight fasting, with holding their breath in maximal expiration in order to minimize the effect of respiration, body position and postprandial changes on the portal flow Endoscopy : Using Sarin classification ( The presence of esophageal varices, their number, exact location, shape, size and cherry-red spots ) Fibroscan: using the standard-probe, and on a fasting (4 h) patient lying flat on his/her back, with the right arm tucked behind the head to facilitate access to the right upper quadrant.

SUMMARY:
The aim of the study is to evaluate the ability of Doppler ultrasonography of the portal vein and liver stiffness measurement using Transient Elestoghraphy in predicting prescence of gastroesophageal variceal and variceal bleeding in patients with liver cirrhosis

DETAILED DESCRIPTION:
Liver cirrhosis incidence and prevalence have been increasing significantly over the years with varying evolutions of etiologies. It is a major cause of mortality and morbidity throughout the world, causing two million deaths per year worldwide (3.5% of all death) with 50% related to cirrhosis complications and 50% related to Hepatocellular Carcinoma and viral hepatitis infections.

Variceal bleeding is among leading causes of death in patients with liver cirrhosis and portal hypertension, In current clinical practice, evaluation of the risk of upper digestive tract bleeding is based on osephagogastroduodenoscopy. Although the occurrence of esophageal varices and the time of gastrointestinal bleeding in portal hypertension cannot be exactly predicted, there are some endoscopic and clinical signs associated with a high risk of bleeding: the size of the esophageal varices, the presence of cherry-red spots (red signs) Recent studies demonstrated that the severity of liver fibrosis, especially the presence of advanced fibrosis defined as stage F3 or F4 fibrosis, is the main driver of prognosis in cirrhosis and the main risk factor for developing not only liver-related events but also extrahepatic complications.

Liver stiffness measurement is a widely used non-invasive tool for the diagnosis of liver fibrosis and has high accuracy, and if combined with platelets count, it can be also used to identify patients at high risk for esophageal varices without the need for endoscopic screening.

Previous studies have demonstrated that liver stiffness can reflect the prognosis of patients with liver cirrhosis because it can indirectly reflect portal hypertension. Liver stiffness measured using transient elastography has been validated as a prognostic quantitative marker for the occurrence of liver-related complications, survival without liver-related death, and overall survival. However, LSM has not been well-verified in the esophageal variceal rebleeding, which is a critical event.

Recent studies indicate also that Doppler ultrasound findings of the portal system and hepatic artery could predict both the presence of varices and the risk of variceal bleeding in patient with portal hypertension and liver cirrhosis.

ELIGIBILITY:
1. Inclusion criteria:

   * Patients > 18 years old.
   * with Liver cirrhosis presented with or without variceal bleeding.
   * or any other complaint, or coming for follow up for their chronic liver disease.
   * with body mass index less than 35.
2. Exclusion criteria:

   * Patients suffering from grade III or grade IV encephalopathy, hepatocellular carcinoma, portal vein thrombosis, and moderate or marked ascites
   * Patients who received drugs that may have a major effect on portal pressure.
   * Patients less than 18 years, patients with BMI more than or equal to 35.
   * pregnant patient.
   * Patients who refused to be involved in our study.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: A case control study will be performed on outpatients and hospitalized patients presented with liver cirrhosis to the department of Tropical medicine, Gastroenterology and Hepatology, Al-Rajhi liver hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
comparing the ability of ultrasound and transient elastography in detecting presence of gastroesoghageal varices to upper endoscopy in liver cirrhosis | baseline
  evaluate the ability of Doppler ultrasonography of the portal vein and liver stiffness measurement using Transient Elestoghraphy in predicting prescence of gastroesophageal varices and variceal bleeding in patients with liver cirrhosis

CONTACTS AND LOCATIONS:
Overall Officials: Hanan Nafeh, professor, Study Director — Vice president of graduate studies of Assiut University

REFERENCES:
- [Background] Plestina S, Pulanic R, Kralik M, Plestina S, Samarzija M. Color Doppler ultrasonography is reliable in assessing the risk of esophageal variceal bleeding in patients with liver cirrhosis. Wien Klin Wochenschr. 2005 Oct;117(19-20):711-7. doi: 10.1007/s00508-005-0424-x. PMID 16416372
- [Background] Xia S, Ren X, Ni Z, Zhan W. A Noninvasive Method-Shear-Wave Elastography Compared With Transient Elastography in Evaluation of Liver Fibrosis in Patients With Chronic Hepatitis B. Ultrasound Q. 2019 Jun;35(2):147-152. doi: 10.1097/RUQ.0000000000000399. PMID 30724863
- See also: Related Info — http://www.frontiersin.org/articles/10.3389/fmed.2021.690825/full